CLINICAL TRIAL: NCT01296165
Title: The Importance of International Travel in the Spread of Extended-spectrum Beta-lactamase-producing Escherichia Coli
Brief Title: International Travel and the Spread of Extended-spectrum Beta-lactamase-producing Escherichia Coli
Status: Completed | Type: Observational
Sponsor: Johann DD Pitout (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Johann DD Pitout, Dr, University of Calgary
Organization: University of Calgary (Other)
Other Study IDs: 38027
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Infection Due to Resistant Bacteria
Keywords: Travel; Spread; Antibiotic resistance

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool specimens
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Travellers visiting India: People that are older than 18 years and planning to visit India for a period of at least 5 days will be approached by the personal at the travel clinics to participate in the study. Informed consent will be obtained prior to enrolling subjects.
  Interventions: Behavioral: Analysing the behaviours of travellers while visiting India

INTERVENTIONS:
Behavioral: Analysing the behaviours of travellers while visiting India — For analyses surrounding the risks for acquisition comparisons between those who acquire ESBLs and those who do not, will be made using Stata version 9.0 (Stata Corp, College Station, TX). Differences in proportions among categorical data will be assessed using Fisher's exact test for pair-wise comparisons. Student T-test or Mann-Whitney U tests will be used for comparing means and medians. For all statistical comparisons a p-value <0.05 will be deemed to represent statistical significance.

SUMMARY:
It is not clear why multi-resistant E. coli (also known as ESBL-producing) have recently became such important causes of infections in patients living and residing in the community. A risk factor analysis study performed during 2004 and 2005 in Calgary had shown that the consumption of the same types of food or well water sources were not significant risk factors for community-associated infections due to these E. coli. However, a significant and unexpected risk factor among these Calgary patients was recent visits to certain high-risk areas such as the Indian subcontinent (India, Pakistan), Africa and the Middle East. Therefore it is possible that international travel to certain high-risk destinations might play, in part, a role in the spread of multi-resistant E. coli across different continents. This would happen via the acquisition of these bacteria in the rectums of returning travelers and the same organism would later cause an infection. However, the evidence that the spread and infections due to ESBL-producing E. coli are associated with international travel is circumstantial at best and the investigators would like to prove that this is indeed true.

The basic idea of the study is to culture the stool of travelers for ESBL-producing E. coli before they leave for India, within seven days after their return to Canada and again after six months. The investigators can then establish which travelers are rectally colonized when visiting India and if these bacteria are still present six months after their return. A detailed questionnaire regarding the traveler's itinerary and behaviours in India will be completed on their return to Canada. The investigators will then compare the itinerary and behaviours of colonized travelers with those of non-colonized travelers and identify certain high-risk behaviours and places for acquiring ESBL-producing E. coli in India. The investigators will also determine if colonized travelers will later develop infections with the same ESBL-producing E. coli they acquired while visiting India.

DETAILED DESCRIPTION:
Title The importance of international travel in the spread of extended-spectrum beta-lactamase-producing Escherichia coli.

Principal investigator Johann DD Pitout, Professor, University of Calgary, Department of Pathology and Laboratory Medicine, no 9, 3535 Research Road NW, Calgary, Alberta, Canada, T2L 2K8. Tel: (403) 770 3338. Fax: (403) 770 3347. johann.pitout@cls.ab.ca

Background and rationale: The changing epidemiology of infections caused by extended-spectrum beta-lactamases-producing bacteria Since 2000 Escherichia coli producing CTX-M enzymes have emerged worldwide as important causes of community-onset urinary tract (UTIs) and blood stream infections due to extended-spectrum beta-lactamase (ESBL)-producing bacteria. Studies from different continents suggested that the sudden worldwide increase of CTX-M-producing E. coli is often due to the emergence of a clone named ST131. It also seems that foreign travel to high-risk areas such as the Indian subcontinent (India, Pakistan) might play, in part, a role in the spread of CTX-M-producing E. coli across different continents. However, the evidence that infections due to ESBL-producing E. coli are associated with international travel is circumstantial and the investigators would like to prove that this is indeed true.

Hypothesis:

Our primary hypothesis is that when travelers visit India, they have a risk of acquiring CTX-M-producing E. coli in their rectums (i.e. there is high risk of rectal colonization with these bacteria). The reason for selecting India is that a previous study from Calgary had shown that the risk for post-travel infections is the highest for travelers returning from this country. The investigators also believe the acquisition of these bacteria is associated with certain high-risk behaviors during travel in India such as drinking water from wells, consuming certain food products or taking antibiotics. Our secondary hypothesis is that some travelers that are colonized with CTX-M-producing E. coli on their return from India, will later develop infections (most likely UITs) with the same bacteria that were first present in their rectums.

Objectives:

To determine the rate of rectal acquisition of ESBL-producing E. coli in travelers to India (i.e. risk of becoming colonized).

To show that same ESBL-producing E. coli persists for up to six months in the rectum of travelers after their return to Canada (i.e. assess the degree of persistence). The investigators suspect that clone ST131 is more likely to be present for longer periods of time than other ESBL-producing E. coli.

To identify the different behaviors of travelers in the India that put them at a high risk for acquiring ESBL-producing E. coli (i.e. risk factors of becoming colonized).

To determine what proportion of colonized travelers will later develop infections with the same ESBL-producing E. coli they acquired while visiting India (i.e. risk of infection).

To characterize the ESBL-producing E. coli and identify clone ST131 among these bacteria.

Study design:

The study will be performed at two travel clinics in Calgary and London, Canada, respectively. These clinics provide comprehensive travel medicine services including preventative vaccinations and prescriptions for anti-malaria drugs. People older than 18 years that are planning to visit India for a period of at least 5 days, will be approached to participate in the study. Informed consent will be obtained prior to enrolling subjects. Travelers who agree to participate will have a detailed travel itinerary and a stool specimen collected prior to travel. Study participants will be requested to return to the travel clinics within 7 days after their return to Canada and complete a detailed questionnaire regarding their behaviors during the visit. The completed questionnaire and stool specimens will be obtained at the second visit. Travelers will be asked to contact the clinics if they develop infections during the next six months. Another stool specimen will be collected six-months after their return to Canada. All stool specimens will be submitted to Calgary Laboratory Services and frozen at -20°C for further analyses. Specimens will be batched and cultured using chromID-ESBL selection media. All ESBL-producing E. coli isolated will undergo phenotypic and genotypic characterization including the identification of clone ST131.

Preliminary data:

During July 2009, 107 stools of patients in Calgary with diarrhea (without a history of recent travel) and 107 of returning travelers with diarrhea, were investigated for the presence of ESBL-producing E. coli; 5/107 (5%) of patients without a history of recent travel had a CTX-M-producing E. coli in their stools while 26/107 (24%) with recent travel were positive for CTX-M-producing E. coli. (p<0.0001). The majority of CTX-Ms were identified as CTX-M-15; 2/5 of the E. coli from the non-travelers belonged to clone ST131 while 6/26 from the travelers belonged to clone ST131.

Statistical methods:

Analyses will be performed using Stata version 9.0 (Stata Corp, College Station, TX). The proportion of patients who become positive will be determined. For further analyses surrounding the risks for acquisition (or subsequent infection), comparisons between those who acquire ESBLs (or get infected) and those who do not, will be made. Differences in proportions among categorical data will be assessed using Fisher's exact test for pair-wise comparisons. Student T-test or Mann-Whitney U tests will be used for comparing means and medians. For all statistical comparisons a p-value <0.05 will be deemed to represent statistical significance.

Overall budget:

The investigators would like to perform the study for a 1-year period and hope to enroll 250 - 300 travelers. The estimated cost is US$250/patient; the overall study cost is US$75000.

ELIGIBILITY:
Inclusion Criteria:

* People that are older than 18 years old
* Planning to visit India for a period of at least 5 days

Exclusion Criteria:

* If a traveler tests positive for ESBL-producing E. coli before leaving for India

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Travelers older than 18 years old that will visit India for longer than 5 days.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To determine the rate of rectal acquisition of ESBL-producing E. coli in travelers to India (i.e. risk of becoming colonized). | 24 months
  Travelers who agree to participate will have a detailed travel itinerary and a stool specimen collected prior to travel. Study participants will be requested to return to the travel clinics within 7 days after their return to Canada and a following-up stool specimen will be obtained at the second visit. The specimens will consist of stool and not rectal swabs. The stool specimens in a transport medium will be submitted to Calgary Laboratory Services and frozen at -20°C for further analyses. The proportion of travelers who become positive for ESBL-producing E. coli will be determined.

SECONDARY OUTCOMES:
To identify the different behaviours of travelers in the India that put them at a high risk for acquiring ESBL-producing E. coli (i.e. risk factors of becoming colonized). | 24 months
  Study participants will be requested to return to the travel clinics within 7 days after their return to Canada and complete a detailed questionnaire regarding their itinerary and behaviours during the visit. The completed questionnaire will be forwarded to the Pitout's laboratory and entered into a central database for further analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Johann Pitout, MD, Principal Investigator — University of Calgary
Locations (1):
- Odessa Travel clinic, Calgary, Alberta, Canada

REFERENCES:
- [Background] Pitout JD, Campbell L, Church DL, Gregson DB, Laupland KB. Molecular characteristics of travel-related extended-spectrum-beta-lactamase-producing Escherichia coli isolates from the Calgary Health Region. Antimicrob Agents Chemother. 2009 Jun;53(6):2539-43. doi: 10.1128/AAC.00061-09. Epub 2009 Apr 13. PMID 19364876
- [Derived] Peirano G, Gregson DB, Kuhn S, Vanderkooi OG, Nobrega DB, Pitout JDD. Rates of colonization with extended-spectrum beta-lactamase-producing Escherichia coli in Canadian travellers returning from South Asia: a cross-sectional assessment. CMAJ Open. 2017 Dec 13;5(4):E850-E855. doi: 10.9778/cmajo.20170041. Epub 2017 Dec 15. PMID 29246886